CLINICAL TRIAL: NCT05740306
Title: Overlap Between Irritable Bowel Syndrome and Celiac Disease - Prospective Survey Study.
Brief Title: Irritable Bowel Syndrome Overlaping Celiac Disease
Acronym: IBSonCD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor
Other Study IDs: 175/2022
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Celiac Disease; Irritable Bowel Syndrome; Overlap Syndrome
Keywords: celiac disease; IBS; overlap syndrome
MeSH Terms: conditions — Celiac Disease; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective observational cohort stuty is to assess the prevalence of overlap irritable bowel syndrome on coeliac disease in patients on gluten-free diet.

The main questions it aims to answer are:

* percentage of the occurrence of irritable bowel syndrome in the population of Polish patients with celiac disease on restrictive gluten-free diet
* what is the correlation between the persistence of intestinal symptoms and adherence to a gluten-free diet (according to the patient's assessment) or confirmation of disease remission (based on histopathology or antibody level).

DETAILED DESCRIPTION:
Based on the data published so far, we plan to assess the occurrence of irritable bowel syndrome symptoms in patients with serologically and histopathologically confirmed celiac disease who follow a gluten-free diet. The assessment will be based on the data collected in the questionnaire published on the website of the Polish Association of People with Celiac Disease and the Gluten Free Diet, while maintaining anonymity and the principles of the GDPR. All patients with celiac disease will be invited to the study, and participation in the survey will be voluntary. The questions included in the survey include demographic, epidemiological and medical data provided by patients and the Rome IV Criteria.

There is no control group or minimum number of participants. The 2nd Department of Gastroenterology has established cooperation with the Board of the Association, which is particularly interested in conducting this type of study and which will be responsible for the technical part of its conduct. The Board of the Association has the powers granted to it by members to contact in scientific matters in the form of mailing and/or posting surveys on the Association's website. We have obtained permission to establish cooperation in this project. The technical department of the website developers will prepare a survey based on the provided templates, which will be placed on the website and/or individual member accounts. Members who have agreed to participate in such health-promoting campaigns will be informed by e-mail. The data obtained back and transferred to the researchers will be anonymized. We assume 12 months time for survey propagation. In the event of recruitment difficulties, the maximum time allowed for recruitment may be 18 months. At this time, we assume a response of about 10% of the members of the association with over 5,500 members.

The disadvantage of the project is the lack of access to patients' medical data to confirm the declared diagnosis and evidence of disease remission, as well as to assess compliance with the diet.

Nevertheless, taking into account that both the assessment of adherence to the diet is a declarative assessment (there are currently no methods of verifying the diet by means of objective indicators) and the criteria for diagnosing IBS are clinical criteria, we believe that the obtained data will allow us to get closer to the problem of overlapping functional diseases.

In addition, the survey does not allow to exclude other organic causes of ailments.

ELIGIBILITY:
Inclusion Criteria:

* serologically and histologically confirmed celiac disease
* informed consent to the study

Exclusion Criteria:

* people who do not follow a gluten-free diet or do not have a diagnosis of celiac disease, but are on a gluten-free diet.

No consent to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with celiac disease who belong to the Polish Association of People with Celiac Disease and the Gluten-Free Diet will be invited to the study, and participation in the survey will be voluntary. There will be a website questionnaire assessing celiac disease diagnosis appropriateness (confirmed histopathologically and present blood antibody) and GFD adherence. Only patients who have confirmed CD and who are on a restrictive diet will be included in the study. The second part of the questionnaire will be addressed irritable bowel syndrome symptoms such as abdominal pain and changes in bowel habits.
  It is worth noticing, that in daily medical practice adherence to the diet is a declarative assessment (there are currently no methods of verifying the diet using objective indicators).
  IBS also is diagnosed only by clinical assessment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
percentage of IBS in CD | one-time answer
  assessment with questionaire the symptoms of irritable bowel syndrome in patients with celiac disease

CONTACTS AND LOCATIONS:
Locations (1):
- Szpital Bielański im. Jerzego Popiełuszki, Warsaw, Masovian Voivodeship, Poland